CLINICAL TRIAL: NCT04533867
Title: Comparison of Palonosetron and Ondansetron for the Prevention of Postoperative Nausea and Vomiting After Bariatric Surgery
Brief Title: Palonosetron vs. Ondansetron for Postoperative Nausea and Vomiting in Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nadir Adnan Hacım, Pirincipal investigator Adnan, Bagcilar Training and Research Hospital
Other Study IDs: Beren Hacım 3
Record Dates: First submitted 2020-08-09; First posted 2020-09-01 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Nausea, Postoperative; Vomiting, Postoperative; Patient Reported Outcomes; Pain, Postoperative; Antiemetics
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Palonosetron; Ondansetron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ondansetron: In Group B (n = 50): Intravenous injection of ondansetron 0.1 mg/kg diluted up to 5 mL with normal saline solution in a maximum dose of 8 mg is performed at the end of bariatric surgery while patients are in anesthesia. The drug is injected once.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy; Drug: Ondansetron 1 mg/kg, max dose 8 mg
- Palonosetron: The antiemetics used are palonosetron in Group A (n = 50): Intravenous injection of Palonosetron 1 mcg/kg diluted up to 5 mL with normal saline solution is performed at the end of bariatric surgery while patients are in anesthesia. The drug is injected once.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy; Drug: Palonosetron 1mcg/kg

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Sleeve gastrectomy, also called a vertical sleeve gastrectomy, is a surgical weight-loss procedure. This procedure is typically performed laparoscopically, which involves inserting small instruments through multiple small incisions in the upper abdomen. During sleeve gastrectomy, about 80 percent of the stomach is removed, leaving a tube-shaped stomach about the size and shape
Drug: Palonosetron 1mcg/kg — Injectable Palonosetron 1 mcg/kg diluted up to 5 mL with normal saline solution and injected intravenously at the end of the bariatric surgery.
  Groups: Palonosetron
Drug: Ondansetron 1 mg/kg, max dose 8 mg — Injectable ondansetron 0.1 mg/kg, maximum of 8 mg was injected intravenously at the end of the bariatric surgery.
  Groups: Ondansetron

SUMMARY:
Evaluate the safety and efficacy of palonosetron versus ondansetron to reduce and control post-operative nausea in bariatric surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is an undesirable clinical condition that increases the likelihood of dehiscence, bleeding, pulmonary aspiration of gastric contents, and electrolyte loss that lead to increased costs, prolonged hospital stays, and delayed recovery. In recent years, selective serotonin 5-hydroxytryptamine sub-type 3 (5-HT3) receptor antagonists such as ondansetron, granisetron, palonosetron have been introduced because they are effective in the prevention and treatment of PONV in bariatric surgery. In this study, the effects of ondansetron and palonosetron on PONV in patients who undergo sleeve gastrectomy will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All morbidity obese patients underwent laparoscopic sleeve gastrectomy

Exclusion Criteria:

drug allergy, intractable nausea and vomiting, gastroesophageal reflux disease, pregnancy, menstruation, the occurrence of nausea or vomiting episodes in the last 24 h prior to surgery, the use of corticosteroids, smoking, alcoholism, the use of psychoactive drugs or any other drug with antiemetic effects, hypersensitivity to other 5-HT3 antagonists, emergency surgeries and chemotherapy within.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — between 18-65 years
Study Population: obese patients underwent laparoscopic sleeve gastrectomy
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Nause and vomiting 6hr | postoperative 6 hours
  Visual Analog Scale score for nausea and vomiting
Nause and vomiting 24hr | postoperative 24 hours
  Visual Analog Scale score for nausea and vomiting
Nause and vomiting 48hr | postoperative 48 hours
  Visual Analog Scale score for nausea and vomiting
Nause and vomiting 72hr | postoperative 72 hours
  Visual Analog Scale score for nausea and vomiting
amount of rescue anti-emetic drugs | postoperative seventh day
  Number of anti emetic metoclopramide intravenous injections during hospitalization and the postoperative one week.

SECONDARY OUTCOMES:
Pain 6hr | postoperative 6 hours
  Visual Analog Scale score for pain
Pain 24hr | postoperative 24 hours
  Visual Analog Scale score for pain
Pain 48hr | postoperative 48 hours
  Visual Analog Scale score for pain
Pain 72hr | postoperative 72 hours
  Visual Analog Scale score for pain

OTHER OUTCOMES:
Functional living index- Emesis | postoperative seventh day
  Quality of life after discharge about emesis using Functional living index- Emesis

CONTACTS AND LOCATIONS:
Overall Officials: Ali Solmaz, Ass. Prof., Study Director — Private Camlıca Erdem Hospital/Istanbul-TURKEY
Locations (2):
- Turkey (Türkiye) (2):
  - Bagcılar Training and Research Hospital, Istanbul
  - Surp Pırgic Armenian Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aydin A, Kacmaz M, Boyaci A. Comparison of ondansetron, tropisetron, and palonosetron for the prevention of postoperative nausea and vomiting after middle ear surgery. Curr Ther Res Clin Exp. 2019 Jun 22;91:17-21. doi: 10.1016/j.curtheres.2019.06.002. eCollection 2019. PMID 31384338
- [Result] Lee S, Kim I, Pyeon T, Lee S, Song J, Rhee J, Jeong S. Population pharmacokinetics of palonosetron and model-based assessment of dosing strategies. J Anesth. 2019 Jun;33(3):381-389. doi: 10.1007/s00540-019-02641-5. Epub 2019 Apr 11. PMID 30976908
- [Result] Rajnikant K, Bhukal I, Kaloria N, Soni SL, Kajal K. Comparison of Palonosetron and Dexamethasone with Ondansetron and Dexamethasone to Prevent Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Cholecystectomy. Anesth Essays Res. 2019 Apr-Jun;13(2):317-322. doi: 10.4103/aer.AER_21_19. PMID 31198253